CLINICAL TRIAL: NCT01321320
Title: Investigation of the Role of FHL-1 and Myostatin in the Development of Intensive Care Unit Acquired Paresis (ICUAP) and the Effect of Increased Muscle Activity on These Pathways.
Brief Title: Investigation of the Role of FHL-1 and Myostatin in Intensive Care Unit Acquired Paresis (ICUAP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government); Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Prof M Polkey, Imperial College London and Royal Brompton Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: CRO1439
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2013-10

CONDITIONS: Intensive Care Unit Acquired Paresis; Muscle Wasting
Keywords: ICUAP; Critical illness; Muscle wasting; ICU
MeSH Terms: conditions — Muscular Atrophy; Critical Illness

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active stimulation (Experimental): This group will receive active muscle stimulation for 1 week to the quadriceps muscle - the leg will be randomly assigned.
  Interventions: Other: Active muscle stimulation

INTERVENTIONS:
Other: Active muscle stimulation — Neuromuscular Electrical stimulation will be applied to one leg (randomly assigned).

SUMMARY:
The primary hypothesis for this study is that Myostatin and FHL-1 are important in the development of ICUAP and that changes in activity levels of muscle will modify the levels of expression and activity of these proteins.

DETAILED DESCRIPTION:
ICUAP is an increasingly recognised clinical problem associated with significant morbidity and mortality. However the pathogenesis of the diseae is poorly understood and as yet no treatment exists. We believe that both myostatin and FHL-1 will be important in the development of this disease. This is based recent research and that both these proteins are likely to be regulated by sepsis and immobility (two major risk factors for ICUAP. There is evidence from invitro work that the two are likely to interact. We have designed an interventional trial to investigate the above hypothesis. Patients admitted to ICU and at risk of developing muscle wasting will be selected and receive electrical muscle stimulation of the quadriceps muscle for 1 week. Physiological measurements of peripheral and respiratory muscle strength and quadriceps size will be made pre and post intervention. And muscle biopsies, blood and urine collected from both legs pre and post intervention. The relevant molecular pathways can then be examined.

ELIGIBILITY:
Inclusion Criteria:

* High risk patients admitted to AICU.

Exclusion Criteria:

* Pre existing neuromuscular disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in muscle myostatin and FHL-1 | 1 week

SECONDARY OUTCOMES:
Change in quadriceps cross sectional area | 1 week
Change in quadriceps strength | 1 week
Change in blood myostatin, miRNA and other markers of muscle breakdown | 1 week
Changes in muscle protein synthesis and breakdown pathways as measured in the muscle biopsy samples. | 1 week
Change in muscle breakdown and synthesis pathways as a factor of amount of muscle stimulation received. | 1 week
Change in muscle phenotype and change in cross sectional area for individual fiber types | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: M Polkey, Principal Investigator — Royal Brompton Hospital and Imperial College; Susannah Bloch, Principal Investigator — Imperial College London
Locations (1):
- National Heart and Lung Institute, Imperial College, London, United Kingdom